CLINICAL TRIAL: NCT04340492
Title: Effectiveness of Adapted Physical Activity Education on Physical Activity Daily in Patients With Parkinson's Disease at an Early Stage
Brief Title: Education for Adapted Physical Activity in Parkinson's Disease
Acronym: ACTIF-PARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018_91; 2019-A02488-49 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Therapeutic Patient Education; Adapted physical activity; Actimetry; Secondary prevention; sensor monitoring
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity group (Experimental)
  Interventions: Other: Education to Adapted Physical Activity
- control group (Sham Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Education to Adapted Physical Activity — 4 group sessions (5 patients) aiming at promoting physical activity, the first three focusing respectively on endurance, posture and balance and power re-enforcement at one-week interval. A fourth session, 3 months latter is a consolidating session aiming at identify and overcome obstacles to practice physical activity in everyday life.
  Arms: Adapted Physical Activity group
Other: Standard care — Standard care concerning Parkinson's disease and physical activity
  Arms: control group

SUMMARY:
Parkinson's disease is a progressive disorders characterized by motor and non-motor symptoms. Actual medical treatments are symptomatic and have little efficacy on late stage axial motor symptoms. Non-pharmacological approaches are therefore essential from the disease onset.

Beside physiotherapy, to practice a regular adapted physical activity is crucial. To implement such a practice in everyday life implies to change habits. Patient Education programs are useful tools to help changing behaviors.

The study evaluate the effect of a program aiming to promote adapted physical activity in early stage Parkinson's disease by comparing patients receiving the program and patients on a waiting list. The hypothesis that the program will increase the one-week mean daily moderate to intense physical activity as measured with an actimeter.

ELIGIBILITY:
Inclusion Criteria:

* suffering from Parkinson's disease according to Movement Disorders Society criteria,
* with a diagnosis of Parkinson for 3 years or less,
* with a stable treatment for Parkinson's disease for 3 months or more,
* having signed the consent form

Exclusion Criteria:

* Woman child-bearing or breath-feeding
* Co-morbidities that influence or contraindicated adapted physical activity (severe respiratory symptoms, cardiopathy…)
* Major depressive disorder according to DSM-V
* Significant cognitive trouble (MOCA<23)
* Atypical parkinson's

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Change in time spent in moderate to vigorous physical activity during one week | between baseline and 6 months after baseline
  Daily physical activity is assessed with an actimeter (Actigraph GT9X).

SECONDARY OUTCOMES:
Change in fatigue as assessed with the Parkinson Fatigue Scale (PFS) | between baseline and 6 months after baseline
  This is a self-evaluation questionnaire, the physical aspects of fatigue and its influence on the everyday functionality and activity. An indication of the presence of clinically relevant fatigue is provided by the mean value calculated from the 16 items. A mean value of > 2.95 indicates the presence of fatigue symptoms
Change in quality of life as assessed with the PDQ-39 scale | between baseline and 6 months after baseline
  Parkinson's Disease Quality of Life Questionnaire (PDQ-39): the 39-Item Parkinson's Disease Questionnaire (PDQ-39) is a commonly used measure of self-appraisal in PD. It is a measure of health status and quality of life, by assessing difficulties in 8 dimensions of daily living: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). The frequency of each event is determined by selecting one of 5 options: never (scored 0) / occasionally (scored 1) / sometimes (2) / often (3) / always (4). Each dimension total score range from 0 to 100, with lower scores reflecting better quality of life.
Change in Non-motor symptoms as assessed with the Non Motor Symptoms Scale (NMSS) | between baseline and 6 months after baseline
  Non-motor symptoms scale for Parkinson's disease (NMSS). Non-motor symptoms are assessed over the last month. Each symptom is scored with respect to:
  Severity: 0 = None; 1 = Mild: symptoms present but causes little distress or disturbance to patient; 2 = Moderate: some distress or disturbance to patient; 3 = Severe: major source of distress or disturbance to patient.
  Frequency: 1 = Rarely (<1/wk); 2 = Often (1/wk); 3 = Frequent (several times per week); 4 = Very Frequent (daily or all the time).
  NMSS contains nine dimensions: cardiovascular (2 items), sleep/fatigue (4 items), mood/cognition (6 items), perceptual problems (3 items), attention/memory (3 items), gastrointestinal (3 items), urinary (3 items), sexual function (2 items), and miscellaneous (4 items).
  Subscores are calculated through multiplication of frequency x severity. Total score is calculated by adding all subscores, range 0-360.
Percentage of patients that complete all four sessions of the program | At 3 months ( duration of the program)
Change in physical activity during one week, assessed with the International Physical Activity Questionnaire (IPAQ) | between baseline and 6 months after baseline
  The International Physical Activity Questionnaire (IPAQ) short form measures walking, moderate- and vigorous intensity, and total PA and daily time spent sitting on weekdays. PA was reported in MET·minutes/week and days per week and was scored using standardized IPAQ scoring protocols to yield total metabolic equivalent minutes (MET·minutes/week) of PA per week. Sitting time was reported as the amount of time in hours and/or minutes participants spent sitting on a weekday during the past seven days.
Change in Motor symptoms as assessed with the MDS-UPDRS-3 | between baseline and 6 months after baseline
  The Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III. MDS-UPDRS Part III measures motor examination. Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0(normal) to 4(severe).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Carriere, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Salengro - Hopital B Chr Lille, Lille, France